CLINICAL TRIAL: NCT04934501
Title: Feasibility of Ultrasound Particle Image Velocimetry to Quantify Flow Near Stented SFA Lesions
Brief Title: Blood Flow Quantification Near Stented SFA Lesions Using Ultrasound Velocimetry
Acronym: EchoPIV in SFA
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-1206
Record Dates: First submitted 2021-06-10; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Computed Tomography Angiography; Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PAD patients: The entire cohort exists of patients recently treated with an endovascular stent placement in the superficial femoral artery (SFA).
  Interventions: Diagnostic Test: High-frame-rate contrast-enhanced ultrasound measurements (echoPIV); Diagnostic Test: Computed tomography angiography (CTA) scan

INTERVENTIONS:
Diagnostic Test: High-frame-rate contrast-enhanced ultrasound measurements (echoPIV) — Patients will undergo high-frame-rate contrast-enhanced ultrasound measurements, within 6 to 8 weeks after the endovascular procedure, at the vascular center of Rijnstate hospital. Prior to these measurements a venous cannula will be placed to ensure venous access for the contrast administration.
Diagnostic Test: Computed tomography angiography (CTA) scan — Patients will undergo a CTA scan of the lower extremities at the Radiology dept. of Rijnstate hospital the same day as the echoPIV measurements. This CTA scan serves as a reference for the vessel geometry and stent location.

SUMMARY:
Peripheral arterial disease (PAD) in the lower extremity is the third leading cause of atherosclerotic cardiovascular morbidity. Endovascular treatment has become the principal surgical strategy in femoro-popliteal lesions. Stent placement induces significant changes in the arterial geometry and thereby in the hemodynamic environment. Visualization of local blood flow patterns (around stents) is challenging, but clinically relevant. Blood flow has a significant influence on the development of atherosclerosis and therefore stent patency. In vivo blood flow characterization might enable the recognition, prediction and explanation of (in-stent) restenosis. This study will therefore aim to investigate the feasibility of a novel ultrasound technique (echoPIV) to quantify spatiotemporal blood flow near stented femoral artery lesions. Furthermore, the blood flow information obtained during the echoPIV measurements will be used as patient-specific boundary conditions in a computational fluid dynamics (CFD) simulation. The tested hypothesis is that blood flow quantification using echoPIV is feasible in and around stents in the femoral artery and that it will improve CFD simulations.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled endovascular treatment of a lesion in the SFA through placement of a bare metal or a covered stent
* A recently (<6 weeks) treated lesion in the SFA through placement of a bare metal or a covered stent

Exclusion Criteria:

* Hypersensitivity to the active substance(s) or any of the excipients in SonoVue
* Right-to-left cardiac shunt
* Severe pulmonary hypertension (pulmonary artery pressure > 90mmHg)
* Uncontrolled systemic hypertension
* Adult respiratory distress syndrome
* Severe pulmonary disease (e.g. COPD GOLD 3/4, adult respiratory distress syndrome)
* Clinically unstable cardiac disease (recent or ongoing myocardial infarction, unstable angina at rest, recent percutaneous coronary intervention, clinically worsening cardiac symptoms, severe cardiac arrythmia's, endocarditis, etc.)
* Prosthetic valves
* Loss of renal function (GFR < 31 ml/min), end-stage renal disease
* End-stage liver disease Sepsis
* Hypercoagulable status, recent thrombosis
* Congestive heart failure (class III or IV)
* Hypersensitivity to iodinated contrast media
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral arterial disease who have been treated with a stent placement in the superficial femoral artery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Qualitative assessment vector velocity fields | 6 to 8 weeks after the procedure (stent placement of SFA)
  Vector velocity fields derived from the echoPIV data will be used to calculate and visualize the velocity profile. In order to answer the question regarding feasibility of echoPIV the quality of the vector velocity fields will be assessed using three different metrics of which the first one is a qualitative assessment by different observers. Recordings of the contrast-enhanced ultrasound with an overlay of the vector velocity profiles will be reviewed on different topics following a scoring rubrics.
Contrast-to-background ratio | 6 to 8 weeks after the procedure (stent placement of SFA)
  The contrast-to-background ratio (CBR) is the second metric to assess the outcomes of the echoPIV measurements. The CBR is a quantitative measure for the contrast levels and therefore for the quality of the contrast-enhanced US image. The higher the CBR level (in dB) the higher the intensity of the contrast which is needed for sufficient PIV analysis.
Vector correlation | 6 to 8 weeks after the procedure (stent placement of SFA)
  The vector correlation is the third metric to assess the outcomes of the echoPIV measurements. The vector correlation demonstrates the tracking performance of the PIV algorithm. The vector correlation provides a unitless value between 0 and 1 in which 0 indicates poor tracking of the microbubble contrast and 1 indicates perfect tracking of the microbubble contrast.

SECONDARY OUTCOMES:
Vorticity | 6 to 8 weeks after the procedure (stent placement of SFA)
  Multiple blood flow parameters will be derived from the echoPIV data. The first one is the vorticity, or the curl of the velocity. The vorticity represents the rotation of particles inside the flow field. This measure can potentially be used to define regions with disturbed blood flow, as a high value (in rad/s) indicates the occurence of a recirculation.
Vector complexity | 6 to 8 weeks after the procedure (stent placement of SFA)
  The second blood flow parameters derived from the echoPIV data is the vector complexity. Vector complexity is a measure of multi-directional flow, ranging from 0 till 1. a value of 1 means complex flow with all velocity vectors pointing in all directions, whereas a value of 0 means laminar flow with all velocity vectors pointing in the same direction. This measure can potentially be used to indicate regions with disturbed blood flow.
Correlation echoPIV and CFD | 6 to 8 weeks after the procedure (stent placement of SFA)
  Velocity profiles obtained with echoPIV will be compared to outcomes of a computational fluid dynamics (CFD) simulation model of the femoral artery. Multiple points along the imaged vessel will be selected in both the echoPIV and the CFD data to extract the temporal velocity profile. This profile will be compared point-by-point after which the correlation between both outcomes/techniques will be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Michel MPJ Reijnen, PhD, Principal Investigator — Dept. of Surgery, Rijnstate Hospital Arnhem
Locations (1):
- Rijnstate Hospital, Arnhem, Gelderland, Netherlands

REFERENCES:
- [Derived] van Helvert M, Engelhard S, Voorneveld J, van der Vee M, Bosch JG, Versluis M, Groot Jebbink E, Reijnen MMPJ. High-frame-rate contrast-enhanced ultrasound particle image velocimetry in patients with a stented superficial femoral artery: a feasibility study. Eur Radiol Exp. 2022 Jul 6;6(1):32. doi: 10.1186/s41747-022-00278-w. PMID 35790584